CLINICAL TRIAL: NCT04663152
Title: Integrated Navigation Services for Treatment Adherence, Counseling, and Research
Acronym: INSTACARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Sonjia Kenya, Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20201234; R01MD018187 (NIH)
Record Dates: First submitted 2020-12-03; First posted 2020-12-10 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: HIV Infection Primary
Keywords: HIV viral suppression; community health worker

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- INSTACARE arm (Experimental): Participants in this arm will receive the INSTACARE intervention for three months.
  Interventions: Behavioral: INSTACARE

INTERVENTIONS:
Behavioral: INSTACARE — CHWs will provide participants with support via phone calls, home-visits, and accompaniment to clinic visits to improve medication management and HIV viral suppression. CHWs will contact participants at least once per week for three months.

SUMMARY:
The goal of this research is to determine whether a Community Health Worker (CHW) intervention including a mobile telehealth (M-Health) component can help achieve long term viral suppression among Black people with poorly controlled HIV.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 years or older
* Miami-Dade Resident at time of enrollment
* self-identify as Black
* Viral load > 200 mL within the last 6-months (VL must be verified via electronic medical record or lab report prior to enrollment)

Exclusion Criteria:

* Any other condition(s) that the treating clinician determines would limit participant from meaningful study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-07-26 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Communication Preferences | 3 months
  Communication preferences will be reported as the number of participants who prefer any of the following intervention modes of administration: text messaging, phone calls, home visits, accompaniment to clinic visits, utilization of existing health portals and phone applications. Data will be collected via survey administered to participants by CHW.
Number of CHW contacts | 3 months
  CHW contacts with participants will be extracted from CHW tracking logs.

CONTACTS AND LOCATIONS:
Overall Officials: Sonjia Kenya, EdD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kenya S, Young B, Escarfuller S, Jones-Weiss D, Carrasquillo O, Riccio A, Yue P. Improving HIV outcomes in Miami's Black populations with clinic-based community health workers protocol: The integrated navigation and support for treatment adherence, counseling, and research (INSTACARE) randomized controlled trial. PLoS One. 2025 Apr 7;20(4):e0316300. doi: 10.1371/journal.pone.0316300. eCollection 2025. PMID 40193336